CLINICAL TRIAL: NCT04573309
Title: A Phase 2, Open-label Study to Assess Copper and Molybdenum Balance in Participants With Wilson Disease Treated With ALXN1840
Brief Title: Copper and Molybdenum Balance in Participants With Wilson Disease Treated With ALXN1840
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1840-WD-204; 2020-001104-41 (EudraCT Number)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Wilson Disease
Keywords: Copper Balance; Molybdenum Balance; Wilson Disease; ALXN1840
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN1840 (Experimental): Participants will be administered ALXN1840 at a dose of 15 milligrams (mg)/day on Day 1 through Day 28 and then increased to 30 mg/day on Day 29 through Day 39
  Interventions: Drug: ALXN1840

INTERVENTIONS:
Drug: ALXN1840 — Administered orally as tablets.
  Other Names: formerly WTX101

SUMMARY:
This exploratory study will investigate the effects of ALXN1840 on copper balance in participants with Wilson disease (WD).

DETAILED DESCRIPTION:
Participants who are treatment experienced (which includes standard-of-care therapies or ALXN1840) and treatment naïve are eligible for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of WD by Leipzig Criteria ≥ 4.
2. Able to reside in the clinical research unit for intensive metabolic monitoring of copper and molybdenum.
3. Participants willing to adhere to copper/molybdenum-controlled diet during the study.
4. Willing and able to follow protocol-specified contraception requirements.
5. Capable of giving signed informed consent.

Exclusion Criteria:

1. Decompensated cirrhosis or model for end stage liver disease score > 13.
2. Modified Nazer score > 7.
3. Clinically significant gastrointestinal bleed within past 3 months.
4. Alanine aminotransferase > 2 × upper limit of normal.
5. Hemoglobin less than lower limit of the reference range for age and sex.
6. Significant medical history (current or past).
7. Previous treatment with zinc within 30 days prior to the Screening Visit.
8. Participants in renal failure, defined as in end-stage renal disease on dialysis (chronic kidney disease stage 5) or creatinine clearance < 30 milliliters/minute.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S. Swenson, MD, PhD, Study Director — Alexion Pharmaceuticals, Inc.; Peter Ksenuk, MD, Study Director — Alexion Pharmaceuticals, Inc.
Locations (3):
- Research Site, New Haven, Connecticut, United States
- Research Site, Grafton, New Zealand
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Participants who had received Wilson disease therapy for >28 days prior to enrollment were administered ALXN1840 at a dose of 15 milligrams (mg)/day on Day 1 through Day 28 and then increased to 30 mg/day on Day 29 through Day 39.
- Cohort 2: Participants who had received Wilson disease therapy for ≤28 days were administered ALXN1840 at a dose of 15 milligrams/day on Day 1 through Day 28 and then increased to 30 mg/day on Day 29 through Day 39.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 8 | 1
Received at Least 1 Dose of Study Drug | 8 | 1
Completed | 7 | 1
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840 treatment.
Groups:
- Cohort 1: Participants who had received Wilson disease therapy for >28 days prior to enrollment were administered ALXN1840 at a dose of 15 mg/day on Day 1 through Day 28 and then increased to 30 mg/day on Day 29 through Day 39.
- Cohort 2: Participants who had received Wilson disease therapy for ≤28 days were administered ALXN1840 at a dose of 15 mg/day on Day 1 through Day 28 and then increased to 30 mg/day on Day 29 through Day 39.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 8 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (12.41) | 26.0 (NA) — NA signfies that standard deviation could not be calculated as there was only 1 evaluable participant. | 34.1 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 7 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Copper Balance: Day 1 Through Day 8
Description: Copper balance is defined as the difference between the measured copper input in food and drink, and the measured copper elimination in urine and feces, and was calculated as the average daily copper balance over the collection period.
Time Frame: Accumulation: Day 1 through Day 8 (ALXN1840 15 mg)
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840 treatment. Here, Number of Participants analyzed signifies those who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams/day | 0.8025 (0.26860) | 0.3062 (NA) — NA signfies that standard deviation could not be calculated as there was only 1 evaluable participant.

2. Secondary Outcome: Change From Baseline In Mean Daily Copper Balance
Description: as for outcome 1
Time Frame: Accumulation: Baseline, Day 1 through Day 8 (ALXN1840 15 mg) and Day 31 through Day 35 (ALXN1840 30 mg); Steady State: Baseline, Day 25 through Day 28 (ALXN1840 15 mg) and Day 36 through Day 39 (ALXN1840 30 mg)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams/day
  Day 1 through Day 8 | -0.3780 (0.14822) | -0.2060 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Day 25 through Day 28 | -0.4697 (0.55770) | 0.1950 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Day 31 through Day 35 | -0.2650 (0.47135) | 0.1492 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Day 36 through Day 39 | -0.1831 (0.44589) | 0.0540 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

3. Secondary Outcome: Copper Quantified In Food, Drink, Feces, And Urine, Including Plasma Total And Labile Bound Copper (LBC)
Description: Copper was assessed through measurement of copper intake (in food and drink), and copper output (in feces and urine) as well as plasma total and labile bound copper.
Time Frame: Accumulation: Day 1 through Day 8 for 15 mg and Day 31 through Day 35 for 30 mg; Steady state: Day 25 through Day 28 for ALXN1840 15 mg and Day 36 through Day 39 for ALXN1840 30 mg
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams
  Copper Food Content: Day 1 through Day 8 | 1.6423 (0.15638) | 1.3523 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Food Content: Day 25 through Day 28 | 1.8269 (0.42485) | 1.5637 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Food Content: Day 31 through Day 35 | 1.8938 (0.21846) | 1.6022 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Food Content: Day 36 through Day 39 | 1.7850 (0.20107) | 1.4397 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Drink Content: Day 1 through Day 8 | 0.0061 (0.00159) | 0.0055 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Drink Content: Day 25 through Day 28 | 0.0066 (0.00180) | 0.0080 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Drink Content: Day 31 through Day 35 | 0.0071 (0.00184) | 0.0044 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Drink Content: Day 36 through Day 39 | 0.0118 (0.00920) | 0.0045 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Feces Content: Day 1 through Day 8 | 0.7594 (0.21993) | 0.7718 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Feces Content: Day 25 through Day 28 | 0.9373 (0.30688) | 0.7238 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Feces Content: Day 31 through Day 35 | 0.8270 (0.33746) | 0.8720 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Feces Content: Day 36 through Day 39 | 0.6136 (0.27213) | 0.7787 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Urine Content: Day 1 through Day 8 | 0.0865 (0.05689) | 0.2798 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Urine Content: Day 25 through Day 28 | 0.1852 (0.09079) | 0.1408 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Urine Content: Day 31 through Day 35 | 0.1584 (0.07823) | 0.0732 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Copper Urine Content: Day 36 through Day 39 | 0.1857 (0.09506) | 0.0994 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

4. Secondary Outcome: Molybdenum Specified In ALXN1840 Doses Given And Quantified In Food, Drink, Feces, And Urine, Including Plasma At Steady State
Description: The amount of molybdenum in food, drink, feces and urine is reported in this outcome measure.
Time Frame: Day 25 through Day 28 (ALXN1840 15 mg) and Day 36 through Day 39 (ALXN1840 30 mg)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams
  Molybdenum Food Content : Days 25 through 28 | 0.3324 (0.18039) | 0.3905 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Food Content : Days 36 through 39 | 0.1923 (0.02354) | 0.1724 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Drink Content : Days 25 through 28 | 0.0006 (0.00012) | 0.0018 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Drink Content : Days 36 through 39 | 0.0007 (0.00024) | 0.0004 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Feces Content : Days 25 through 28 | 1.1004 (0.38506) | 1.0656 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Feces Content : Days 36 through 39 | 1.0541 (0.83207) | 2.1352 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Days 25 through 28 | 0.7250 (0.32736) | 0.5480 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Days 36 through 39 | 0.8984 (0.62633) | 1.0395 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

5. Secondary Outcome: Change From Baseline In Total Molybdenum Excretion In Urine And Feces
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams
  Molybdenum Feces Content : Day 1 through 8 | 0.7102 (0.22072) | 0.9510 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Feces Content : Days 25 through 28 | 1.0146 (0.42658) | 0.9736 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Feces Content : Days 31 through 35 | 1.0484 (0.62291) | 1.7188 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Feces Content : Days 36 through 39 | 0.9683 (0.88027) | 2.0432 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Day 1 through 8 | 0.3972 (0.15972) | 0.1725 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Days 25 through 28 | 0.6122 (0.28154) | 0.4010 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Days 31 through 35 | 0.7974 (0.47607) | 0.8085 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Molybdenum Urine Content : Days 36 through 39 | 0.7855 (0.58820) | 0.8926 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

6. Secondary Outcome: Mean Daily Molybdenum Balance At ALXN1840 Steady State
Description: Molybdenum balance at steady state was assessed through measurement of molybdenum intake (in food, drink, and ALXN1840), and molybdenum output (in feces and urine). Steady state is defined as molybdenum (out) equal to molybdenum (in).
Time Frame: Steady state: Day 25 through Day 28 (ALXN1840 15 mg) and Day 36 through Day 39 (ALXN1840 30 mg)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams/day
  Days 25 through 28 | 1.3618 (0.44254) | 2.1087 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Days 36 through 39 | 2.7599 (1.68008) | 3.6581 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

7. Secondary Outcome: Accumulation Of Molybdenum As Determined By Molybdenum Balance
Description: Molybdenum balance was assessed through measurement of molybdenum intake (in food, drink, and ALXN1840), and molybdenum output (in feces and urine).
Time Frame: Accumulation: Day 1 through Day 8 (ALXN1840 15 mg) and Day 31 through Day 35 ((ALXN1840 30 mg)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
milligrams
  Days 1 through 8 | 2.2458 (0.23232) | 2.0876 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.
  Days 31 through 35 | 2.6265 (1.96365) | 4.0775 (NA) — NA signifies that standard deviation could not be calculated as there was only 1 evaluable participant.

8. Primary Outcome: Mean Daily Copper Balance: Day 31 Through Day 35
Description: as for outcome 1
Time Frame: Accumulation: Day 31 through Day 35 (ALXN1840 30 mg)
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840 treatment.
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 1
milligrams/day | 0.9156 (0.37982) | 0.6613 (NA) — NA signfies that standard deviation could not be calculated as there was only 1 evaluable participant.

9. Primary Outcome: Mean Daily Copper Balance: Day 25 Through Day 28
Description: as for outcome 1
Time Frame: Accumulation: Day 25 through Day 28 (ALXN1840 15 mg)
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840 treatment.
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 1
milligrams/day | 0.7109 (0.67915) | 0.7072 (NA) — NA signfies that standard deviation could not be calculated as there was only 1 evaluable participant.

10. Primary Outcome: Mean Daily Copper Balance: Day 36 Through Day 39
Description: as for outcome 1
Time Frame: Accumulation: Day 36 through Day 39 (ALXN1840 30 mg)
Population: Full analysis set included all participants who received at least 1 dose of ALXN1840 treatment.
Measure: Mean (Standard Deviation); unit: milligrams/day
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 8 | 1
milligrams/day | 0.9975 (0.26543) | 0.5662 (NA) — NA signfies that standard deviation could not be calculated as there was only 1 evaluable participant.

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Total Molybdenum and Plasma Ultrafiltrate (PUF) Molybdenum
Time Frame: Day 1 up to Day 39
Population: Pharmacokinetic (PK) analysis set included all participants who had sufficient plasma samples to enable the calculation of PK parameters and provide PK profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliters
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 7 | 1
nanograms/milliliters
  Total Molydenum | 430.451 (46.6) | 1271.551 (NA) — NA signifies that Geometric Coefficient of Variation (CV) could not be calculated as there was only 1 evaluable participant.
  Plasma ultrafiltrate molybdenum | 13.546 (43.5) | 17.823 (NA) — NA signifies that geometric CV could not be calculated as there was only 1 evaluable participant.

12. Secondary Outcome: Area Under The Concentration Time Curve (AUC0-inf) of Total Molybdenum and Plasma Ultrafiltrate (PUF) Molybdenum
Time Frame: Day 39
Population: Pharmacokinetic analysis set included all participants who had sufficient plasma samples to enable the calculation of PK parameters and provide PK profiles. Here, Number of participants analyzed signifies those who were evaluable for this outcome measure and number analyzed signifies those who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliters
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 1
hours*nanograms/milliliters
  Total Molydenum | 13532.591 (49.3) | 65694.679 (NA) — NA signifies that geometric CV could not be calculated as there was only 1 evaluable participant.
  Plasma ultrafiltrate molybdenum: number analyzed (Participants) | 5 | 1
  Plasma ultrafiltrate molybdenum | 292.737 (11.9) | 476.960 (NA) — NA signifies that geometric CV could not be calculated as there was only 1 evaluable participant.

ADVERSE EVENTS:
Time Frame: Baseline up to Day 56
Description: Safety set included all participants who received at least 1 dose of ALXN1840.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 6/8 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT04573309/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT04573309/SAP_001.pdf